CLINICAL TRIAL: NCT05487729
Title: Low Back Pain Prevalence in Young Adults.
Brief Title: Low Back Pain Prevalence
Acronym: LBP_TRA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: LBP_TRA
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain; Local Stabilizers; ODI
Keywords: low back pain; local stabilizers; ODI
MeSH Terms: conditions — Low Back Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults: Young adults without neurological and serious structural condition.
  Interventions: Other: ultrasonography and functional assessment and questionnaire survey

INTERVENTIONS:
Other: ultrasonography and functional assessment and questionnaire survey — ultrasonography and functional assessment and questionnaire survey

SUMMARY:
Brief Summery: Low back pain is a significant, serious and widespread problem in our world today, both in terms of social and economic burdens. It should be emphasized that even the young adult age group is very often affected by non-specific, low back pain without proven pathoanatomical changes.

The aim of our current study is to assess the prevalence of low back pain among young adults, and we would like to examine the musculoskeletal and psychosocial factors associated with low back pain that can be justified as risk factors. Our further goal is to assess and compare lumbar sensorimotor control in young people without complaints and with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* in case of patients with low back pain: chronic pain
* in case of asymptomatic individuals: no symptomes

Exclusion Criteria:

* serious neurologycal symptomes
* serious scoliosis
* previous surgery which affected the local stabilizers
* serious pulmonar disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female, male, other
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-08-08 (Estimated); Study Completion 2024-05-08 (Estimated)

PRIMARY OUTCOMES:
DIAGNOSTICAL ULTRASOUND - MUSCULOSKELETAL ULTRASOUND | 12 minutes
  An imaging procedure that allows doctors, physiotherapist to see muscles, joints, and more. For diagnosing muscle tears/strains, nerves, and arthritis. Physical therapy or injection of medicine may be next step. Involves radiology and center for musculoskeletal care.
NEUROCOM BASIC BALANCE MASTER | 20 minutes
  Limits of Stability (LOS), Modified Clinical Test of Sensory Interaction on Balance (mCTSIB), Rhythmic Weight Shift (RWS) special tests for the balancing and motor control paremeters.
STABILIZER PRESSURE BIOFEEDBACK | 5 minutes
  Stabilizer Pressure Biofeedback is an easy to use device that provides a visual indication of whether you are working the correct postural muscles, in the right manner, when performing specific exercises. Intended for the prevention and treatment of back pain, neck pain, and to improve core stability
ZEBRIS CMS-10 ULTRASOUND SYSTEM | 10 minutes
  ZEBRIS CMS10 computer-controlled, ultrasound-based motion analysis system located in the Biomechanical Laboratorium
The Functional Movement Screen (FMS) | 10 minutes
  The Functional Movement Screen (FMS) is a screening tool used to evaluate seven fundamental movement patterns in individuals with no current pain complaint or musculoskeletal injury. The FMS is not intended to diagnose orthopedic problems but rather to demonstrate opportunities for improved movement in individuals. The screen is designed to place an individual in extreme positions where movement deficits become noticeable if appropriate stability and mobility are not used.
STABILITY LIMIT TESTS | 12 minutes
  LATERAL REACH, MODIFIED LATERAL REACH, REACH FORWARD, MODIFIED REACH FORWARD: special functional tests for stability limit.

SECONDARY OUTCOMES:
VISUAL ANALOG SCALE | 1 minute
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. VAS is the most common pain scale.
MEDICAL HISTORY RECORD SHEET | 3 minutes
  We created an individual patient examination form, in which we could ask our subjects about their lifestyle habits and about their low back pain.
OSWESTRY DISABILITY INDEX | 3 minutes
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.
ROLAND-MORRIS QUESTIONNAIRE | 2 minutes
  The Roland-Morris Disability Questionnaire[1] is designed to assess self-rated physical disability caused by low back pain. The Roland-Morris Disability Questionnaire is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain.
THE QUEBEC BACK PAIN DISABILITY SCALE (QBPDS) | 2 minutes
  The Quebec back pain disability scale is a condition-specific questionnaire developed to measure the level of functional disability for patients with low back pain (LBP) is a condition-specific questionnaire developed to measure the level of functional disability for patients with low back pain (LBP). The original purpose of the questionnaire is to take into account the functional limitations related to pain, to monitor the progress of individual patients and to compare the evolution of LBP subjects incorporated in rehabilitation programs.
SHORT FORM-36 HEALTH SURVEY | 4 minutes
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.
THE STATE-TRAIT ANXIETY INVENTORY (STAI Y-1,2 form)) | 4 minutes
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress
THE PERCEIVED STRESS SCALE (PSS) | 2 minutes
  The Perceived Stress Scale is a classic stress assessment instrument. The tool remains a popular choice for helping us understand how different situations affect our feelings and our perceived stress. The questions in this scale ask about your feelings and thoughts during the last month. In each case, you will be asked to indicate how often you felt or thought a certainn way.
THE BECK DEPRESSION INVENTORY (BDI, BDI-1A, BDI-II) | 4 minutes
  It is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Its development marked a shift among mental health professionals, who had until then, viewed depression from a psychodynamic perspective, instead of it being rooted in the patient's own thoughts.
  There are three versions of the BDI-the original BDI, first published in 1961 and later revised in 1978 as the BDI-1A, and the BDI-II, published in 1996. The BDI is widely used as an assessment tool by health care professionals and researchers in a variety of settings.
LOW BACK PAIN KNOWLEDGE QUESTIONNAIRE (LKQ) | 2 minutes
  This instrument assesses knowledge about back pain. Composed of 16 questions, divided into the following categories: general aspects, concepts and treatment. The score ranges from 0 to 24 points, with a higher score denoting a better knowledge of low back pain.
COMI | 2 minutes
  The COMI is a valid and sensitive questionnaire for the evaluation of patients with degenerative lumbar disease before and after treatment. The COMI is a questionnaire composed of 8 questions that evaluates pain (2 items), function (1 item), well-being (1 item), disability (2 items) and satisfaction (2 items). The scores of the questionnaire range from 1 to 5, with 1 being the best possible result. The total COMI score is the average of the 5 dimensions. It was designed for a simpler but effective standardized evaluation of outcome in patients with low back pain and would replace more cumbersome health-related questionnaires in daily practice.
ZUNG | 1 minute
  The Zung Self-Rating Depression Scale was designed by W.W. Zung to assess the level of depression for patients diagnosed with depressive disorder. The Zung Self-Rating Depression Scale is a short self-administered survey to quantify the depressed status of a patient. There are 20 items on the scale that rate the four common characteristics of depression: the pervasive effect, the physiological equivalents, other disturbances, and psychomotor activities. There are ten positively worded and ten negatively worded questions. Each question is scored on a scale of 1-4 (a little of the time, some of the time, good part of the time, most of the time).
PISQ-IR | 2 minutes
  PISQ-IR is a disease-specific questionnaire to assess sexual function in women with pelvic floor disorders.
FSFI | 3 minutes
  The Female Sexual Function Index (FSFI) is recognized as an excellent tool for assessing female sexuality and screening female sexual dysfunction, but it also has important venereological implications as sexually transmitted diseases result from human behaviour in the sexual sphere.
GAUDENZ | 2 minutes
  The Gaudenz Incontinence Questionnaire has been used widely in Europe as a diagnostic tool to discriminate between SUI and UUI. Initial studies demonstrated high validity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Csongrád-Csanád, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kasza BB, Nakity K, Finta R, Pasztor N, Kurokawa T, Sapi M, Domjan A. Investigating the impact of perceived stress and anxiety on nonspecific low back pain among future health care professionals in Hungary: a cross-sectional study. Front Psychol. 2025 May 19;16:1463414. doi: 10.3389/fpsyg.2025.1463414. eCollection 2025. PMID 40458634